CLINICAL TRIAL: NCT00694746
Title: Randomized Trial of Fish Oil Versus Placebo to Reduce ALT Levels in Overweight Adolescents
Brief Title: Study of Fish Oil to Reduce ALT Levels in Adolescents
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed for slow recruitment
Sponsor: Boston University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Carine Lenders, Carine Lenders, MD, MS, ScD, Boston University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIT40
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Non-alcoholic Fatty Liver Disease; Fatty Liver
Keywords: ALT; Non-Alcoholic Fatty Liver Disease; Adolescents; Overweight; Treatment
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Overweight | interventions — Omacor; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Experimental): Omega-3-acid ethyl esters in the form of fish oil capsules with ram up from 1g to 4 g/day (capsules 1g)
  Interventions: Drug: Omega-3-acid ethyl esters
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3-acid ethyl esters — Participants will receive 2 capsules of 1 gram of fish oil with meals twice a day for a period of six months (including a ramp up period of three weeks)
  Other Names: Omacor; Lovaza
  Arms: Fish oil
Drug: Placebo — Participants will receive 2 capsules of 1 gram of placebo with meals twice a day for a period of six months (including a ramp up period of three weeks)
  Other Names: corn oil
  Arms: Placebo

SUMMARY:
This trial will provide preliminary data to test the hypothesis that a six-month treatment period with fish oil for overweight adolescent with mild to moderate persistent elevation of ALT levels and presence of hepatic steatosis on CT-scan is safe and will result in decreased ALT.

DETAILED DESCRIPTION:
Over the past two decades, pre-adult nonalcoholic fatty liver disease (NAFLD) has emerged from the relative obscurity to become the most common cause of liver disease in pediatric patients. Currently, over 17% of US children and adolescents have a BMI at or greater than the 95th percentile for age and gender and 20% of children in weight management programs are estimated to have NAFLD. Untreated NAFLD can lead to fibrosis and to established cirrhosis in children as young as 10. Fish oils are a rich source of omega-3-acid ethyl esters or n-3 long-chain polyunsaturated fatty acids, and increasing evidence suggest they may safely improve hepatic steatosis. Given the prevalence of obesity, of NAFLD, and the severe, progressive nature of this condition, effective treatment strategies are urgently needed. We plan to gather preliminary data on the efficacy and safety of fish oil supplements in reducing persistent elevation of ALT levels and hepatic steatosis on abdominal CT-scan among urban youth (BMI>=95th percentile). This preliminary data will provide the necessary information to calculate the sample size for a phase 2 trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI (kg/m2) at or above the 95th percentile for age and gender
* Weight below 400 pounds (less than 182 kilograms)
* Persistent elevation of ALT (41-90 UI/L at study screening)
* Presence of hepatic steatosis on abdominal CT-scan
* Able to give informed consent/assent

Exclusion Criteria:

* Type 2 diabetes mellitus
* Prior drug treatment for diabetes, insulin insensitivity, or weight loss medications six months before screening
* Use of prescription strength glucocorticoids within three months before screening
* History of syndrome or medical disorder associated with significant obesity
* Participation in a weight loss program within six months of screening resulting in 5% or more weight loss
* History of weight loss surgery
* Alcohol use more than twice weekly or more than 3 alcohol containing beverages within a 24-hour period in the past six months
* Known or suspected bleeding condition
* History of liver disease including prior liver biopsy with NASH type 2 or cirrhosis
* Former or present positive blood tests for Infectious hepatitis B or C, autoimmune hepatitis, Wilson disease, Alpha-1 anti-trypsin deficiency, Iron storage disease, or high TSH
* History of past or current pregnancy
* Use of illegal/illicit drugs
* Other conditions contraindicated or cause for caution in the use of fish oil
* Unable to comply with the protocol
* Any other serious disease determined by the study gastroenterologists and physician nutrition specialist as potential study risk for the patient

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Efficacy parameters: Characterize the reduction in ALT levels. | 3 and 6 months from baseline
Safety/compliance parameters: Describe the safety blood tests results, review of systems, and physical examination at baseline, mid point, and end of treatment, as well as identify adverse events and compliance parameters at study contacts. | From baseline to end of treatment

SECONDARY OUTCOMES:
Improvement in waist circumference, insulin and lipid indices, and other metabolic parameters. | 3 and 6 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Carine M Lenders, MD, MS, ScD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Design with difficult enrollement